CLINICAL TRIAL: NCT01445678
Title: A Multicenter, Double-Blind, Randomized, Phase 3 Study to Compare the Efficacy and Safety of Intravenous CXA-201 With That of Meropenem in Complicated Intraabdominal Infections
Brief Title: Study Comparing the Safety and Efficacy of Intravenous CXA-201 and Intravenous Meropenem in Complicated Intraabdominal Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7625A-004; CXA-cIAI-10-09 (Other: Cubist Study Number); CXA-cIAI-10-08 (Other: Cubist Study number for 7625A-003); NCT01445665 (obsolete NCT alias)
Record Dates: First submitted 2011-09-26; First posted 2011-10-04 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Complicated Intra-abdominal Infection
Keywords: cIAI
MeSH Terms: interventions — Metronidazole; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CXA-201 and Metronidazole as treatment for cIAI (Experimental)
  Interventions: Drug: CXA-201 and metronidazole
- Meropenem as treatment for cIAI (Active Comparator)
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: CXA-201 and metronidazole — CXA-201 IV infusion (1500mg q8h) and metronidazole IV infusion (500mg q 8h) for 4-14 days
  Arms: CXA-201 and Metronidazole as treatment for cIAI
Drug: Meropenem — Meropenem IV infusion (1000mg q8h) for 4-14 days
  Arms: Meropenem as treatment for cIAI

SUMMARY:
This is a Phase 3, multicenter, prospective, randomized, double-blind, double dummy study of CXA-201 Intravenous (IV) infusions (1500mg q8h) and metronidazole (500mg q8h) versus meropenem (1000mg q8h)for the treatment of adults with Complicated Intraabdominal Infections (cIAI).

DETAILED DESCRIPTION:
Approximately, 500 subjects will be enrolled into this study, randomized 1:1 to receive CXA-201 and metronidazole or comparator (meropenem). Subject participation will require a minimum commitment of 38 days and a maximum of 45 days. An End of Treatment (EOT) visit will occur within 24 hours following the last dose of study drug administration/drug discontinuation. A Test of Cure (TOC)/Safety visit will be conducted 26 to 30 days following the first dose of study drug administration. A Last Follow-up (LFU) visit will be conducted 38 to 45 days after the first dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of cIAI.
* Subject requires surgical intervention (e.g., laparotomy, laparoscopic surgery, or percutaneous draining of an abscess) within 24 hours of (before or after) the first dose of study drug.

Exclusion Criteria:

* Simple appendicitis; acute suppurative cholangitis; infected necrotizing pancreatitis; pancreatic abscess; or pelvic infections.
* Complicated intraabdominal infection managed by staged abdominal repair (STAR), open abdomen technique including temporary closure of the abdomen, or any situation where infection source control is not likely to be achieved.
* Use of systemic antibiotic therapy for IAI for more than 24 hours prior to the first dose of study drug, unless there is a documented treatment failure with such therapy.
* Have a concomitant infection at the time of randomization, which requires non-study systemic antibacterial therapy in addition to IV study drug therapy. (Drugs with only gram-positive activity [e.g., daptomycin, vancomycin, linezolid] are allowed).
* Severe impairment of renal function (estimated CrCl < 30 mL/min), or requirement for peritoneal dialysis, hemodialysis or hemofiltration, or oliguria (< 20 mL/h urine output over 24 hours).
* The presence of hepatic disease at baseline.
* Considered unlikely to survive the 4 to 5 week study period.
* Any rapidly-progressing disease or immediately life-threatening illness (including respiratory failure and septic shock).
* Have a documented history of any moderate or severe hypersensitivity or allergic reaction to any β-lactam antibacterial (a history of a mild rash followed by uneventful re-exposure is not a contraindication to enrollment), including cephalosporins, carbapenems, penicillins, or ß-lactamase inhibitors, or metronidazole, or nitroimidazole derivatives.
* Women who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2011-12-23 (Actual); Primary Completion 2013-10-03 (Actual); Study Completion 2013-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Hershberger, Pharm.D, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (61):
- United States (4):
  - Springfield, Illinois
  - Boston, Massachusetts
  - Robbinsdale, Minnesota
  - Columbus, Ohio
- Argentina (12):
  - Ciudadelo-Buenos Aires, Buenos Aires
  - General Rodríguez, Buenos Aires
  - La Plata, Buenos Aires
  - Loma Hermosa, Buenos Aires
  - Luján, Buenos Aires
  - Merlo, Buenos Aires
  - Tandil, Buenos Aires
  - Vicente López, Buenos Aires
  - Paraná, Entre Ríos Province
  - Corrientes
  - Córdoba
  - Santa Fe
- Bulgaria (3):
  - Pleven
  - Sofia
  - Varna
- Chile (2):
  - Temuco, Cautin
  - Santiago
- Croatia (2):
  - Split, Dalmatia
  - Zagreb
- Estonia (3):
  - Kohtla-Järve
  - Tallinn
  - Tartu
- Germany (2):
  - Freiburg im Breisgau, Baden-Weurttemberg
  - Heidelberg, Baden-Wurttemberg
- Hungary (9):
  - Gyula, Bekes County
  - Szeged, Csongrád megye
  - Szentes, Csongrád megye
  - Győr, Győr-Moson-Sopron
  - Zalaegerszerg, Zala County
  - Budapest
  - Kaposvár
  - Kecskemét
  - Vác
- Israel (4):
  - Kfar Saba, Sharon
  - Tel Litwinsky, Tel Aviv
  - Beer Yahkov
  - Haifa
- Latvia (2):
  - Liepāja
  - Riga
- Lithuania (4):
  - Kaunas
  - Klaipėda
  - Šiauliai
  - Vilnius
- Chisinau, Moldova
- Poland (5):
  - Krakow, Lesser Poland Voivodeship
  - Lubin, Lublin Voivodeship
  - Wołomin, Masovian Voivodeship
  - Szczecin, West Pomeranian Voivodeship
  - Lodz, Łódź Voivodeship
- Serbia (4):
  - Belgrade
  - Krafujevac
  - Niš
  - Novi Sad
- South Korea (4):
  - Wŏnju, Gangwon-do
  - Incheon, Gyeonggi-do
  - Suwon, Gyeonggi-do
  - Seoul

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Popejoy MW, Long J, Huntington JA. Analysis of patients with diabetes and complicated intra-abdominal infection or complicated urinary tract infection in phase 3 trials of ceftolozane/tazobactam. BMC Infect Dis. 2017 May 2;17(1):316. doi: 10.1186/s12879-017-2414-9. PMID 28464828
- [Derived] Xiao Y, Tong ML, Liu LL, Lin LR, Chen MJ, Zhang HL, Zheng WH, Li SL, Lin HL, Lin ZF, Xing HQ, Niu JJ, Yang TC. Novel predictors of neurosyphilis among HIV-negative syphilis patients with neurological symptoms: an observational study. BMC Infect Dis. 2017 Apr 26;17(1):310. doi: 10.1186/s12879-017-2339-3. PMID 28446129
- [Derived] Kullar R, Wagenlehner FM, Popejoy MW, Long J, Yu B, Goldstein EJ. Does moderate renal impairment affect clinical outcomes in complicated intra-abdominal and complicated urinary tract infections? Analysis of two randomized controlled trials with ceftolozane/tazobactam. J Antimicrob Chemother. 2017 Mar 1;72(3):900-905. doi: 10.1093/jac/dkw486. PMID 27999024
- [Derived] Miller B, Popejoy MW, Hershberger E, Steenbergen JN, Alverdy J. Characteristics and Outcomes of Complicated Intra-abdominal Infections Involving Pseudomonas aeruginosa from a Randomized, Double-Blind, Phase 3 Ceftolozane-Tazobactam Study. Antimicrob Agents Chemother. 2016 Jun 20;60(7):4387-90. doi: 10.1128/AAC.03074-15. Print 2016 Jul. PMID 27139477
- [Derived] Solomkin J, Hershberger E, Miller B, Popejoy M, Friedland I, Steenbergen J, Yoon M, Collins S, Yuan G, Barie PS, Eckmann C. Ceftolozane/Tazobactam Plus Metronidazole for Complicated Intra-abdominal Infections in an Era of Multidrug Resistance: Results From a Randomized, Double-Blind, Phase 3 Trial (ASPECT-cIAI). Clin Infect Dis. 2015 May 15;60(10):1462-71. doi: 10.1093/cid/civ097. Epub 2015 Feb 10. PMID 25670823

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two identical P3 protocols were initiated (NCT01445678 and NCT01445665) subsequently, Cubist and FDA agreed that integrated data from the 2 protocols could be analyzed and reported in a single Clinical Study Report. A total of 993 subjects were randomized to both arms, 493 to NCT5678 and 500 to NCT5665. Of these, 485 and 494 received treatment.
Groups:
- CXA-201 and Metronidazole as Treatment for cIAI: CXA-201 and metronidazole: CXA-201 IV infusion (1500mg q8h) and metronidazole IV infusion (500mg q 8h) for 4-14 days.
  Of the 979 treated subjects in the integrated analysis set, 482 received CXA.
- Meropenem as Treatment for cIAI: Meropenem: Meropenem IV infusion (1000mg q8h) for 4-14 days Of the 979 treated subjects in the integrated analysis set, 497 received meropenem.
Period: Overall Study
Arm/Group | CXA-201 and Metronidazole as Treatment for cIAI | Meropenem as Treatment for cIAI
Started | 482 | 497
Completed | 452 | 476
Not Completed | 30 | 21
Not completed — Adverse Event | 12 | 8
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 8 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CXA-201 and Metronidazole as Treatment for cIAI | Meropenem as Treatment for cIAI | Total
Number analyzed (Participants) | 482 | 497 | 979
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (17.94) | 50.5 (16.85) | 50.5 (17.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 195 | 401
  Male | 276 | 302 | 578

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects With Clinical Outcome of Cure at the Test of Cure (TOC) Visit in the Microbiological Intent to Treat (MITT) Population
Description: Clinical cure is complete resolution or significant improvement in signs and symptoms of the index infection, such that no additional antibacterial therapy or surgical or drainage procedure was required for the index infection.
Time Frame: TOC; 26-30 days after start of study drug administration
Population: MITT: Randomized patients, with baseline pathogen.
Measure: Number; unit: percentage of subjects
Arm/Group | CXA-201 and Metronidazole as Treatment for cIAI | Meropenem as Treatment for cIAI
Number analyzed (Participants) | 389 | 417
percentage of subjects | 83.0 | 87.3
Statistical Analysis 1: Comparison: CXA-201 and Metronidazole as Treatment for cIAI vs Meropenem as Treatment for cIAI; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the lower bound of the 2-sided 95% confidence interval was greater than -10%; Risk Difference (RD) = -4.2, 95% CI 2-sided [-8.91 to 0.54]

2. Secondary Outcome: The Percentage of Subjects With Microbiological Outcome of Success at the TOC Visit in the Microbiologically Evaluable (ME) Population
Description: Success is eradication (absence of the baseline pathogen in a specimen appropriately obtained from the original site of infection) or presumed eradication (absence of material to culture in a subject who was assessed as a clinical cure) for each baseline pathogen
Time Frame: TOC; 26-30 days after start of study drug administration
Population: Microbiologically evaluable: Treated patients, complied with protocol, with pathogens susceptible to study drug.
Measure: Number; unit: percentage of subjects
Arm/Group | CXA-201 and Metronidazole as Treatment for cIAI | Meropenem as Treatment for cIAI
Number analyzed (Participants) | 275 | 321
percentage of subjects | 94.2 | 94.7
Statistical Analysis 1: Comparison: CXA-201 and Metronidazole as Treatment for cIAI vs Meropenem as Treatment for cIAI; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the lower bound of the 2-sided 95% confidence interval was greater than -10%; Risk Difference (RD) = -1.0, 95% CI 2-sided [-4.52 to 2.59]

3. Secondary Outcome: The Percentage of Subjects With Clinical Response at End of Therapy (EOT) Visit in the MITT Population
Description: Clinical response is complete resolution or significant improvement in signs and symptoms of the index infection, such that no additional antibacterial therapy or surgical or drainage procedure was required for the index infection.
Time Frame: EOT; Within 24 hours of last study drug administration
Population: MITT: Microbiological Intent-to-Treat: Randomized patients, with baseline pathogen.
Measure: Number; unit: percentage of subjects
Arm/Group | CXA-201 and Metronidazole as Treatment for cIAI | Meropenem as Treatment for cIAI
Number analyzed (Participants) | 389 | 417
percentage of subjects | 89.2 | 92.3
Statistical Analysis 1: Comparison: CXA-201 and Metronidazole as Treatment for cIAI vs Meropenem as Treatment for cIAI; Test type: Superiority or Other; Risk Difference (RD) = -3.1, 95% CI 2-sided [-7.23 to 0.89]

4. Secondary Outcome: The Percentage of Subjects With Clinical Response at End of Therapy in the ME Population
Description: as for outcome 3
Time Frame: EOT; Within 24 hours of last study drug administration
Population: Microbiologically evaluable: Treated patients, complied with protocol, with pathogens susceptible to study drug.
Measure: Number; unit: percentage of subjects
Arm/Group | CXA-201 and Metronidazole as Treatment for cIAI | Meropenem as Treatment for cIAI
Number analyzed (Participants) | 275 | 321
percentage of subjects | 97.1 | 97.5
Statistical Analysis 1: Comparison: CXA-201 and Metronidazole as Treatment for cIAI vs Meropenem as Treatment for cIAI; Test type: Superiority or Other; Risk Difference (RD) = -0.4, 95% CI 2-sided [-3.4 to 2.33]

5. Secondary Outcome: The Percentage of Subjects With Clinical Response at Long Term Follow-Up (LFU) in the MITT Population
Description: Clinical response is clinical cure at TOC and no signs and symptoms recur or worsen since the TOC visit.
Time Frame: LFU; 38 to 45 days after first study drug administration
Population: MITT: Randomized patients, with baseline pathogen.
Measure: Number; unit: percentage of subjects
Arm/Group | CXA-201 and Metronidazole as Treatment for cIAI | Meropenem as Treatment for cIAI
Number analyzed (Participants) | 389 | 417
percentage of subjects | 82.5 | 86.6
Statistical Analysis 1: Comparison: CXA-201 and Metronidazole as Treatment for cIAI vs Meropenem as Treatment for cIAI; Test type: Superiority or Other; Risk Difference (RD) = -4.1, 95% CI 2-sided [-9.09 to 0.94]

6. Secondary Outcome: The Percentage of Subjects With Clinical Response at LFU Visit in the ME Population
Description: Clinical response is clinical cure at TOC and no signs and symptoms recur or worsen since the TOC visit
Time Frame: LFU; 38 to 45 days after first study drug administration
Population: Microbiologically evaluable: Treated patients, complied with protocol, with pathogens susceptible to study drug.
Measure: Number; unit: percentage of subjects
Arm/Group | CXA-201 and Metronidazole as Treatment for cIAI | Meropenem as Treatment for cIAI
Number analyzed (Participants) | 258 | 304
percentage of subjects | 100 | 99.3
Statistical Analysis 1: Comparison: CXA-201 and Metronidazole as Treatment for cIAI vs Meropenem as Treatment for cIAI; Test type: Superiority or Other; Risk Difference (RD) = 0.7, 95% CI 2-sided [-0.88 to 2.37]

ADVERSE EVENTS:
Arm/Group | CXA-201 and Metronidazole as Treatment for cIAI | Meropenem as Treatment for cIAI
Serious Adverse Events (participants affected / at risk) | 39/482 | 36/497
Other Adverse Events (participants affected / at risk) | 159/482 | 138/497
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CXA-201 and Metronidazole as Treatment for cIAI (N=482) | Meropenem as Treatment for cIAI (N=497)
Septic shock (Infections and infestations) | 3 | 2
Abdominal abscess (Infections and infestations) | 2 | 2
Pelvic abscess (Infections and infestations) | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Adominal infection (Infections and infestations) | 1 | 0
Infectious peritonitis (Infections and infestations) | 1 | 0
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 0 | 2
Subdiaphragmatic abscess (Infections and infestations) | 0 | 2
Appendiceal abscess (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Gallbladder abscess (Infections and infestations) | 0 | 1
Graft infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 2 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Multi-organ failure (General disorders) | 3 | 0
Sudden death (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Intra-abdominal haemorrhage (Vascular disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Transient ischaemic attach (Nervous system disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Bilary fistula (Hepatobiliary disorders) | 0 | 1
Perforation bile duct (Hepatobiliary disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CXA-201 and Metronidazole as Treatment for cIAI (N=482) | Meropenem as Treatment for cIAI (N=497)
Anaemia (Blood and lymphatic system disorders) | 6 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 8 | 5
Atrial fibrillation (Cardiac disorders) | 6 | 2
Tachycardia (Cardiac disorders) | 7 | 9
Abdominal pain (Gastrointestinal disorders) | 6 | 2
Constipation (Gastrointestinal disorders) | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 30 | 25
Dyspepsia (Gastrointestinal disorders) | 2 | 7
Nausea (Gastrointestinal disorders) | 37 | 28
Vomiting (Gastrointestinal disorders) | 16 | 19
Oedema peripheral (General disorders) | 9 | 4
Pyrexia (General disorders) | 25 | 20
Pneumonia (Infections and infestations) | 5 | 4
Anaemia postoperative (Injury, poisoning and procedural complications) | 9 | 8
Seroma (Injury, poisoning and procedural complications) | 6 | 7
Alanine aminotransferase increased (Investigations) | 7 | 5
Aspartate aminotransferase increased (Investigations) | 5 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 14 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 3
Dizziness (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 12 | 9
Anxiety (Psychiatric disorders) | 9 | 7
Insomnia (Psychiatric disorders) | 17 | 11
Dysuria (Renal and urinary disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Rash (Skin and subcutaneous tissue disorders) | 4 | 5
Hypertension (Vascular disorders) | 9 | 10
Hypotension (Vascular disorders) | 8 | 4
Phlebitis (Vascular disorders) | 2 | 5

LIMITATIONS AND CAVEATS:
Two identical P3 protocols were initiated (NCT01445678 and NCT01445665) subsequently, Cubist and FDA agreed that integrated data from the 2 protocols could be analyzed and reported in a single Clinical Study Report. These analyses are presented here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator(s) must undertake not to submit any part of the data from this protocol for publication without the prior consent of Cubist Pharmaceuticals, Inc.